CLINICAL TRIAL: NCT04715828
Title: Impact of Ionizing Treatment on the Nuclear Structure of Human Spermatozoa.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020 PONS-REJRAJI
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Sperm Preservation; Irradiated Semen
Keywords: Fertility Preservation; Ionizing radiation; Human sperm; Thyroid Cancer; Nuclear alterations; Telomere length; DNA Fragmentation and Oxidation; Chromatin decondensation; Conventional sperm parameters
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- control arm "fresh": Fresh semen treated without irradiation before cryopreservation
  Interventions: Other: Cryopreserved semen
- control arm "cryopreserved": cryopreserved semen without irradiation (n=60)
  Interventions: Other: Cryopreserved semen
- acute irradiation at low dose: Pelvis scanning : acute irradiation (1 or 2 second) using low dose (n=30),
  Interventions: Other: Acute and low irradiation
- long irradiation at low dose: Bone scintigraphy : long irradiation (3h) using low dose (n=30),
  Interventions: Other: Long and low irradiation
- long irradiation at medium dose: Radioactive Iodine 131 therapy (RAT) applied for thyroid cancer : long irradiation (3h) using medium dose (n=60),
  Interventions: Other: Long and medium irradiation

INTERVENTIONS:
Other: Cryopreserved semen — sperm will be frozen in Cryosperm® cryoprotectant medium (Origio). The samples will be packaged in previously identified high security straws (Cryobiosystem). Slow freezing of the straws will be carried out using the Nanodigicool® programmable device (Cryobiosystem).
  Groups: control arm "cryopreserved"; control arm "fresh"
Other: Acute and low irradiation — sperm sample will be placed on the scanner's processing table to be exposed for 1 to 2 seconds. Several dose levels will then be made in order to limit the value of 17 mGy
  Groups: acute irradiation at low dose
Other: Long and low irradiation — sperm sample will be exposed to gamma radiation by adding a solution of Tc99m for 3 hours.
  Groups: long irradiation at low dose
Other: Long and medium irradiation — sperm sample will be exposed to gamma radiation by adding a solution of I131 for 3 hours
  Groups: long irradiation at medium dose

SUMMARY:
Differentiated thyroid cancer is the third cause of cancer in young men of childbearing age. Its treatment by irradiation with Radioactive Iodine 131 therapy (RAT) could alter spermatogenesis and result in azoospermia and permanent infertility. A preventive gametes cryopreservation was recommended before RAT, but without mentioning a period of teratogenic risk transmissible to the offspring. To date, RAT impact on human sperm nucleus is poorly known or even unknown, notably on telomere length.

Our objective is to define RAT effects on human sperm nucleus by in vitro irradiation exposure of human spermatozoa to mimicking that of the gonads in the context of irradiation with iodine131 used for thyroid cancer. We will analyze standard sperm parameters, major DNA alterations and telomere length using molecular and cellular assays. Nucleus morphology and chromatin organization will also be analyzed using 3D bio-imaging. This study will permit to optimize the indications for the preservation of fertility.

DETAILED DESCRIPTION:
Our main objective is to measure the in vitro impact of irradiation treatment on sperm nuclear quality such as DNA fragmentation and oxidation, chromatin condensation and organisation, nucleus morphology and notably sperm telomere length (STL).

The secondary objectives are :

* to measure RAT impact on sperm parameters (vitality, motility and morphology)
* to measure the impact of cryopreservation on chromatin organisation and nucleus morphology
* to evaluate RAT impact on human sperm cells in comparison with cryopreservation
* to evaluate the impact of different doses and types of irradiation on human sperm cells
* to establish relations between potential alterations of standards sperm parameters (vitality, motility and morphology) and nuclear sperm parameters (DNA fragmentation and oxidation, chromatin condensation and organisation, nucleus morphology and STL.

Our final goal is to provide a significant improvement of men fertility diagnosis and optimize our fertility preservation practices.

To this end, we will expose ejaculated human spermatozoa (n = 90) at different (low and moderate) doses of gamma or X photons to mimic gonads irradiation. Absorbed doses by the samples were calculated using the GATE Monte Carlo platform (version 8.2). Experiment geometry settings were modelled as three dimension voxelized volumes inside the software by assigning a shape, size, distance and density for all the volumes created. All measurements will be made on surplus samples from men undergoing routine semen analysis at the Center for Reproductive Medicine, after receiving their written informed consent. Semen samples are collected and subdivided into 3 arms to analyse sperm quality after:

* irradiation exposure (3 conditions);
* a freezing- thawing cycle;
* fresh state: negative control without treatment.

Before (fresh state) and after each treatment we will analyse:

* standard semen parameters (vitality, motility and morphology) in accordance with WHO, 2010;
* STL using Flow FISH, q-PCR and q-FISH;
* chromatin condensation (chromomycin A3);
* DNA oxidization (8-OHdG residues);
* DNA fragmentation (TUNEL);
* 3D nucleus structure using 3D bio-imaging.

ELIGIBILITY:
Inclusion Criteria:

* Man less than 45 years
* Man undergoing routine semen analysis at the Center for Reproductive Medicine, accepting the research protocol and signing the associated consent will be included in the protocol without distinction of physical criteria.

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: All measurements are made on surplus samples from men undergoing routine semen analysis at the Center for Reproductive Medicine, after receiving their written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
To measure in vitro the impact of an ionizing radiation treatment on sperm nuclear quality and in particular the size of telomeres. | 01/01/2018-01/01/2022
  To achieve this goal, we will expose human sperm to an irradiation dose of I131 to mimic the irradiation of gonads and sperm. Reliquat of semen will be cryopreserved (control condition). After thawing, the same sample will be subdivised into 2 groups in order to analyze the sperm quality :
  * After an irradiation dose of I131
  * After a cryopreservation

SECONDARY OUTCOMES:
To measure in vitro the impact of an irradiation dose of I131 on sperm nuclear quality, notably on STL. | 01/01/2018-01/01/2022
  All measurements are made on surplus samples from men undergoing routine semen analysis at the Center for Reproductive Medicine, after receiving their written informed consent. Semen samples will be collected and subdivided into 3 arms to analyse sperm quality after:
  * irradiation exposure (3 conditions);
  * a freezing- thawing cycle;
  * fresh state: negative control without treatment.
  Before (fresh state) and after each treatment we will analyse:
  * STL using Flow FISH, q-PCR and q-FISH;
  * chromatin condensation (chromomycin A3);
  * DNA oxidization (8-OHdG residues);
  * DNA fragmentation (TUNEL);
  * 3D nucleus structure using 3D bio-imaging.
to measure RAT impact on sperm parameters (vitality, motility and morphology) | 01/01/2018-01/01/2022
  All measurements are made on surplus samples from men undergoing routine semen analysis at the Center for Reproductive Medicine, after receiving their written informed consent. Semen samples will be collected and subdivided into 3 arms to analyse sperm quality after:
  * irradiation exposure (3 conditions);
  * a freezing- thawing cycle;
  * fresh state: negative control without treatment.
  * a freezing- thawing cycle;
  * fresh state: negative control without treatment. Before (fresh state) and after each treatment we will analyse standard semen parameters (vitality, motility and morphology) in accordance with WHO, 2010;
To measure in vitro the impact of cryopreservation on sperm nuclear quality, notably on STL, chromatin organisation and nucleus morphology | 01/01/2018-01/01/2022
  All measurements are made on surplus samples from men undergoing routine semen analysis at the Center for Reproductive Medicine, after receiving their written informed consent. Semen samples will be collected and subdivided into 3 arms to analyse sperm quality after:
  * irradiation exposure (3 conditions);
  * a freezing- thawing cycle;
  * fresh state: negative control without treatment.
  Before (fresh state) and after each treatment we will analyse:
  * STL using Flow FISH, q-PCR and q-FISH;
  * chromatin condensation (chromomycin A3);
  * DNA oxidization (8-OHdG residues);
  * DNA fragmentation (TUNEL);
  * 3D nucleus structure using 3D bio-imaging.
to evaluate RAT impact on human sperm cells in comparison with cryopreservation | 01/01/2018-01/01/2022
  We will compare effects induced by RAT and cryopreservation on each sperm sample. In order to limit the bias, for each irradiation treatment, a sample of sperm cells (cryopreserved control) will be treated under identical conditions.
to evaluate the impact of different doses and types of irradiation on human sperm cells | 01/01/2018-01/01/2022
  All measurements are made on surplus samples from men undergoing routine semen analysis at the Center for Reproductive Medicine, after receiving their written informed consent. Semen samples will be collected and subdivided into 3 arms to analyse sperm quality after:
  * irradiation exposure (3 conditions);
  * a freezing- thawing cycle;
  * fresh state: negative control without treatment.
  Irradiation exposure will be realised under 3 conditions:
  * acute and low irradiation : sperm sample will be placed on the scanner's processing table to be exposed for 1 to 2 seconds. Several dose levels will then be made in order to limit the value of 17 mGy.
  * long and low irradiation: sperm sample will be exposed to gamma radiation by adding a solution of Tc99m for 3 hours.
  * long and medium irradiation : sperm sample will be exposed to gamma radiation by adding a solution of I131 for 3 hours
to establish relations between potential alterations of standards sperm parameters (vitality, motility and morphology) and nuclear sperm parameters (DNA fragmentation and oxidation, chromatin condensation and organisation, nucleus morphology and STL. | 01/01/2018-01/01/2022
  We will correlate the effects induced by on vitality, motility and morphology and nuclear sperm parameters (DNA fragmentation and oxidation, chromatin condensation and organisation, nucleus morphology and STL.

CONTACTS AND LOCATIONS:
Overall Officials: Hanae PONS-REJRAJI, PhD, Study Chair — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided